CLINICAL TRIAL: NCT03713476
Title: Effectiveness of a Robot Assisted Tenodeis-grip Neurorehabilitation for Upper Extremity Function of Stroke Patients
Brief Title: Effectiveness of a Robot Assisted Tenodeis-grip Neurorehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-BR-106-074-T
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-03

CONDITIONS: Rehabilitation, Tenodesis, Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted training (Experimental): The participants will receive 20 minutes of robot assisted tenodesis-grip therapy, followed by 20 minutes of regular motor task specific training in each treatment session.
  Interventions: Other: Motor task training
- Traditional occupational therapy (Active Comparator): The participants will receive 20 minutes of traditional occupational therapy (sensorimotor facilitation techniques, such as: Rood, Bobath and propriocetive-neuromuscular-facilitation), followed by 20 minutes of motor task specific training in each treatment session.
  Interventions: Other: Motor task training

INTERVENTIONS:
Other: Motor task training — motor task specific training

SUMMARY:
In the proposed study, the investigators assumed that using robot assisted tenodesis-grip training providing high does assisted grip movement may do the effects on motor shaping and greater brain priming for hand paresis of the stroke patients. The specific aim of this study is to examine the difference in the treatment effects between the combination of robot assisted tenodesis-grip training with task-oriented training and combination of traditional occupational therapy with task-oriented training on the motor, sensation, hand performance of the stroke patients. The expected outcomes of this research are to help the clinicians understand the training mechanism and effects of robot assisted tenodesis-grip training on functional performance of upper extremity for unilateral stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of stroke with unilateral side involved;
2. Stroke at least 7 days before the start of the first assessment session;
3. A score of Mini-mental state examination greater than 24 for proving higher mental function;
4. Premorbid right-handedness.

Exclusion Criteria:

1. Uncontrolled hypertension;
2. Major cognitive-perceptual deficit;
3. Other brain disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Change in the result of Fugl-Meyer assessment for UE motor function | baseline, 6 weeks and 18 weeks
  Each item is rated on a three-point ordinal scale (2 points for the detail being performed completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.
Change in the result of Modified Ashworth scale (MAS) | baseline, 6 weeks and 18 weeks
  Muscle tone is defined by the resistance of a muscle being stretched without resistance.
Change in the result of Box and blocks test | baseline, 6 weeks and 18 weeks
  The score is the number of blocks carried from one box to the other in one minute. Higher values represent a better outcome.
Change in the result of Semmes-Weinstein monofilament (SWM) test | baseline, 6 weeks and 18 weeks
  The Semmes-Weinstein monofilamenttest examines the cutaneous pressure threshold, range from 1.65-6.65. Higher values represent a worse outcome.
Change in the result of Motor Activity Log | baseline, 6 weeks and 18 weeks
  MAL is a structured interview with testing sensitivity used to examine how much (amount of use, AOU) and how well (quality of movement, QOM) the subject uses their more-affected arm. For the 30 items MAL, each item is scored on a 0-5-ordinal scale.

SECONDARY OUTCOMES:
Clinical global impression scale | post-intervention (week 6)
  Self-reported improvement over the treatment period,. The scale, rated from 1 (very much improved) to 7 (very much worse), is as the indicator for determining perceptible change of the patients for assisted tenodeis-grip robot system.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Hsu HY, Koh CL, Yang KC, Lin YC, Hsu CH, Su FC, Kuo LC. Effects of an assist-as-needed equipped Tenodesis-Induced-Grip Exoskeleton Robot (TIGER) on upper limb function in patients with chronic stroke. J Neuroeng Rehabil. 2024 Jan 3;21(1):5. doi: 10.1186/s12984-023-01298-2. PMID 38173006
- [Derived] Hsu HY, Yang KC, Yeh CH, Lin YC, Lin KR, Su FC, Kuo LC. A Tenodesis-Induced-Grip exoskeleton robot (TIGER) for assisting upper extremity functions in stroke patients: a randomized control study. Disabil Rehabil. 2022 Nov;44(23):7078-7086. doi: 10.1080/09638288.2021.1980915. Epub 2021 Sep 29. PMID 34586927